CLINICAL TRIAL: NCT05259631
Title: Inhalational (Sevoflurane) Versus Intravenous (Propofol) Sedation in Adults With a Moderate Form of ARDS: A Multicentral Randomized Pilot Trial
Brief Title: Inhalational (Sevoflurane) Versus Intravenous (Propofol) Sedation in Adults With a Moderate Form of ARDS
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Financial problems
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, Head of the Research V. Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INVERSE
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Sedation; Sevoflurane; Propofol; Volatile anesthetics; Intravenous anesthetics; Inhalational anesthetics; Intensive care unit
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhalational sedation (Experimental)
  Interventions: Drug: Sevoflurane
- Intravenous sedation (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Patients are to be sedated by sevoflurane inhalation. For this purpose, any certificated devices are suitable - AnaConDa or Mirus evenly. Starting dose of sevoflurane is to be 2 ml/h and may be modified at the discretion of the attending intensivist to achieve and maintain the target level of sedation
  Arms: Inhalational sedation
Drug: Propofol — Patients of this group will receive an intravenous infusion of propofol with starting dose of 1 mg/kg/h. The precise dose to maintain the desired level of sedation is left at the discretion of the attending intensivist and may be revised at any time. The upper dose limit for propofol is 4 mg/kg/h. In case of tolerance to propofol infusion, midazolam or antipsychotics (haloperidol) can be added to achieve the desired level of sedation
  Arms: Intravenous sedation

SUMMARY:
The American European Consensus Conference (AECC) 1994 defined acute respiratory distress syndrome (ARDS) as an acute inflammatory syndrome manifesting as diffuse pulmonary edema and respiratory failure that cannot be explained by, but may co-exist with, left-sided heart failure. During the sequel Conference of the European Society of Intensive Care Medicine, in 2012 minor changes were made, and since that so-called Berlin definition of ARDS is used worldwide for the description of this severe disease. Three grades of severity were proposed to distinguish ARDS according to the level of hypoxemia with a mortality of 24% in patients with mild ARDS, rising to 48% in those with severe ones.

Systemic inflammation is considered to be the main reason of ARDS. Activated neutrophils interact with the alveolar-capillary membrane causing the increasing permeability with the sequence lung edema's development. Inflammatory exudate inactivates surfactant leading to collapse and consolidation of distal airspaces with progressive loss of the lung's gas exchange surface area. Unfortunately, systemic inflammatory response syndrome (SIRS) simultaneously inhibits the mechanism of active pulmonary vasoconstriction and allows deoxygenated blood to pass through unventilated areas of the lung boosting the right-to-left shunt. Both mechanisms lead to hypoxemia, which is the main and obligatory feature of ARDS.

Actually, endothelial dysfunction and transcapillary leakage seem to be one of the main steps in the development of respiratory failure during ARDS. Last decades it was found out that glycocalyx is also participating in this process too.

Thus, it became clear that substances preserving endothelium and glycocalyx from SIRS-causing damage may have a beneficial effect in ARDS treatment. It seems to be crucially important so as the majority of drugs failed to demonstrate any positive effects in terms of ARDS treatment.

To the moment we have some evidence, which came from experimental studies, that halogenated anesthetics can preserve glycocalyx against ischemia-reperfusion injury.

The primary objective for the multicentral INVERSE Trial will be to determine the effects of inhalational (sevoflurane) versus intravenous (propofol) sedation on P/F ratio on the second day, hospital mortality and ICU (intensive care unit), and in-hospital length of stay in adults with a moderate form of ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Endotracheal intubation or tracheostomy
* Timing: Acute onset of new or worsening of chronic respiratory symptoms within 72 hours before the randomization
* Chest imaging: Bilateral opacities-not fully explained by effusions, lobar/lung collapse, or nodules
* Origin of edema: Respiratory failure not fully explained by cardiac failure or fluid overload
* Oxygenation: 100 mm Hg < PaO2/FiO2 ≤ 200 mm Hg with PEEP ≥ 5 cm H2O

Exclusion Criteria:

* History or family history of malignant hyperthermia
* History of propofol infusion syndrome
* Documented or suspected increased intracranial pressure
* Chronic restrictive pulmonary disease
* Chronic obstructive pulmonary disease
* Neuromuscular disease
* Chest wall disorder
* Pulmonary vascular disease
* NYHA class ≥ 3
* Severe pulmonary hypertension (mean pulmonary artery pressure > 40 mmHg)
* Documented ongoing COVID-19 infection
* Ongoing immunosuppressive therapy
* Previous randomization in this trial
* Post randomization exclusion criterion: Documented ongoing COVID-19 infection during the first 48 hours after the randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
P/F ratio | day 2 after the randomization
  PaO2 divided on FiO2

SECONDARY OUTCOMES:
28-days mortality | 28 day
  number of deaths
6-months mortality | 6 months
  number of deaths
1-year mortality | 1 year
  number of death
Length of stay in the intensive care unit | 1 year
  number of days in the intensive care unit
Length of hospitalization | 1 year
  number of days in hospital
Ventilator free days in ICU | 1 year
  number of days in ICU - number of days on mechanical ventilation
Ventilator free days during hospitalization | 1 year
  Length of hospitalization - number of days on mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, Principal Investigator — Negovsky Reanimatology Research Institute
Locations (1):
- Demikhov Municipal Clinical Hospital 68, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No